CLINICAL TRIAL: NCT03873701
Title: Bedside Ultrasonography in Acute Patients With Suspected Kidney Involvement
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Pernilla Goldberg Borggaard, BSc med, Odense University Hospital
Other Study IDs: 65004
Record Dates: First submitted 2018-10-30; First posted 2019-03-13 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Hydronephrosis; Pyelonephritis; Urosepsis
Keywords: bedside ultrasonography; emergency department
MeSH Terms: conditions — Hydronephrosis; Pyelonephritis; Emergencies | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: bedside ultrasonography — Patients suspicious to urinary tract infection with kidney involvement are being examined by ultrasonography to detect hydroneprhosis. The treating clinicians fill out questionnaires to validate the impact of the bedside ultrasonography on the patient care and treatment.
  Other Names: Ultrasound

SUMMARY:
The aim of this study is to evaluate the accuracy and implications of the diagnoses and treatment determined by bedside ultrasonography (b-US) of the kidneys compared to current clinical assessment. Potentially diagnosing patients faster and avoiding missing conditions leading to readmission or unnecessary radiation from computed tomography (CT).

This study evaluates the use of b-US as a supplement to clinical evaluation, in an unselected group of patients in the emergency department (ED) with signs of kidney involvement. The b-US of the kidneys is performed by a medical student certified in this technique. The evaluation will be based on data collected from a Danish hospital (Odense University Hospital, OUH) in autumn 2018.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of urinary tract infection and one or more of the following:
* Flank pain
* Fever
* Symptoms when voiding
* Creatinine elevation or 20% elevation from known creatinine level elevation

Exclusion Criteria:

* Age < 18 years
* Radiological ultrasonographic examination already performed
* Patients who are not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single-center population collected from patients with contact to the emergency department (ED) at Odense University Hospital (OUH). Convenience sample.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic hydronephrosis | All included patient undergo bedside ultrasonography within 4 hours after admission
  Ultrasonographic hydronephrosis defined by > 1cm pelvic dilation

SECONDARY OUTCOMES:
Clinical consequence of bedside ultrasonographic result | Within 4 hours after admission
  Clinicians responsible for the primary clinical assessment determine treatment and further examinations before and after the ultrasonographic results.

CONTACTS AND LOCATIONS:
Overall Officials: Annmarie T Lassen, Professor, Study Director — Forskningsenheden FAM OUH
Locations (1):
- Odense Universitetshospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No